CLINICAL TRIAL: NCT03242954
Title: Innovative Approaches for Minor Consent: Consent 2.0 - A Multi-Center Study of the Adolescent Medicine Trials Network for HIV/AIDS Interventions (ATN)
Brief Title: Innovative Approaches for Minor Consent: Consent 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Amelia Knopf, Assistance Professor, IU School of Nursing, Indiana University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-0538; 5U24HD089880-02 (NIH)
Record Dates: First submitted 2017-08-03; First posted 2017-08-08 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-03

CONDITIONS: HIV

STUDY DESIGN:
Intervention Model Description: Consent 2.0 has a parallel group-like design for adolescents. Adolescents will be randomized into 1 of 3 consent conditions using a randomized block design that is stratified by study site and the adolescent's natal sex. The order in which the hypothetical trials are presented to adolescents will be randomized using a block design. A subset of 6-8 adolescents per site will be selected for a debriefing interview.
  Consent 2.0 has a crossover-like design for parents. Parents will provide feedback on all three consent conditions and for both hypothetical trials. The order in which the hypothetical trials are presented to parents will be determined using a randomized block design that is stratified by study site and the parent's adolescent's natal sex. The presentation order for the 3 consent condition vignettes for each hypothetical trial will be determined using a randomized block design. A subset of 6-8 parents by site will be selected for debriefing interview.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adolescents: Consent Condition 1 (Active Comparator): Autonomous minor consent
  Interventions: Other: Autonomous minor consent
- Adolescents: Consent Condition 2 (Active Comparator): Adult permission required
  Interventions: Other: Adult permission required
- Adolescents: Consent Condition 3 (Active Comparator): Parental permission required
  Interventions: Other: Parental permission required
- Parents: Consent Conditions 1-3 (Active Comparator): Autonomous minor consent, adult permission required, and parental permission required
  Interventions: Other: Autonomous minor consent; Other: Adult permission required; Other: Parental permission required

INTERVENTIONS:
Other: Autonomous minor consent — Consent requirement where the participant is not required to get anyone's permission to participate in the trial.
  Arms: Adolescents: Consent Condition 1; Parents: Consent Conditions 1-3
Other: Adult permission required — Consent requirement where the participant is required to obtain an adult's permission to participate in the trial.
  Arms: Adolescents: Consent Condition 2; Parents: Consent Conditions 1-3
Other: Parental permission required — Consent requirement where the participant is required to obtain their parent's permission to participate in the trial.
  Arms: Adolescents: Consent Condition 3; Parents: Consent Conditions 1-3

SUMMARY:
The purpose of this study is to examine how the consent process affects the acceptability of participation in biomedical HIV prevention trials, from the perspective of behaviorally high-risk minors and the parents of minor adolescents.

DETAILED DESCRIPTION:
Potential participants will be recruited from clinical settings and HIV testing centers. If interested in participation, they will take a short Computer Assisted Self-Interview (CASI) screening survey to determine eligibility. Those eligible will take part in the one-day study visit at that time or will provide contact information to set up the study visit at a later date.

All study participants will attend a one-day study visit at their respective study site. Upon arrival, participants will complete a CASI that collects demographic, social, behavioral, and attitudinal measures. Next, participants will take part in a simulated consent process for two hypothetical trials modeled after ATN 113 and HPTN 077. Study procedures differ for adolescents and parents, so each group is described separately below:

Adolescent Participants: For each hypothetical trial, research staff will lead the participant through a simulated consent process consistent with their randomized consent condition. Then, the participant will complete a CASI assessing Willingness to Participate (WTP) and will work with research staff to complete the University of San Diego (UCSD) Brief Assessment of Capacity to Consent (UBACC).

Parent Participants: For each hypothetical trial, research staff will review the informed consent forms with the parent. The parent will complete a CASI with three vignettes that describe each of the three possible consent conditions. Parents will rate the acceptability of each vignette. Then, the participant will work with research staff to complete the UCSD Brief Assessment of Capacity to Consent (UBACC). Finally, the participant will answer a series of questions via CASI.

A subset of 6-8 adolescents and 6-8 parents per study site will complete a debriefing interview assessing adolescent and parent perspectives on the various consent conditions in greater depth, and to better understand the role of study features, family, and adolescent characteristics in willingness to participate/willingness to support the hypothetical research studies.

ELIGIBILITY:
Note: Age limits apply to adolescent participants and to the adolescent children of parent participants.

Adolescent Inclusion Criteria

* Age 14-17 inclusive
* Able to read and speak English
* HIV status is negative or unknown
* Engaged in high-risk sexual activity in the last six months

Adolescent Exclusion Criteria

* Child of a parent already enrolled in the study

Parent Inclusion Criteria

* Able to read and speak English
* Parent or guardian of an adolescent who is between ages 14-17
* The parent/guardian's adolescent's HIV status is either negative or unknown

Parent Exclusion Criteria

* Parent of a child already enrolled in the study

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 254 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2019-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Knopf, PhD, MPH, RN, Principal Investigator — Indiana University School of Medicine; Matthew Psioda, PhD, Study Director — University of North Carolina, Chapel Hill
Locations (4):
- United States (4):
  - Children's Hospital Colorado/Univ of Colorado SOM, Aurora, Colorado
  - University of South Florida, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University/SOM, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: Yes
De-identified study data will be made available in the NICHD Data and Specimen Hub (DASH), a centralized resource for researchers to store de-identified data from NICHD supported studies for use in secondary research. NICHD DASH is a free public resource designed for the scientific research community.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available after data analyses have been completed, data has been de-identified, and all DASH submission requirements have been met and approved. Data will be available according to NICHD DASH timelines.
Access Criteria: Please see DASH guidelines for access criteria.
URL: https://dash.nichd.nih.gov/

REFERENCES:
- [Derived] Knopf A, Draucker CB, Fortenberry JD, Ott MA, Arrington-Sanders R, Reirden D, Schneider J, Straub D, Ofner S, Bakoyannis G, Zimet G. Parental Engagement in Consent Processes for Enrollment in Biomedical HIV Prevention Trials: Implications for Minor Adolescents' Willingness to Participate. J Adolesc Health. 2023 May;72(5):703-711. doi: 10.1016/j.jadohealth.2022.11.241. Epub 2023 Jan 14. PMID 36646563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 1,366 individuals were screened at 4 study sites in the United States (Chicago, Denver, Baltimore, and Tampa) between May 2018 and September 2019. Of those screened, 422 met all eligibility criteria and 254 were randomized, enrolled, and completed the 1-time study visit.
Pre-assignment Details: All parent participants are considered one study 'arm' as they were not randomized to just one of the three consent conditions (as the adolescent participants were), but rather were presented with information on all 3 consent conditions and commented on the acceptability of each.
Groups:
- Adolescents: Consent Condition 1: Autonomous consent
  Autonomous consent: Consent requirement where the participant is not required to get anyone's permission to participate in the trial.
- Parents: Consent Conditions 1-3: Autonomous consent, Adult permission required and Parental permission required
  Autonomous consent: Consent requirement where the participant is not required to get anyone's permission to participate in the trial.
  Adult permission required: Consent requirement where the participant is required to obtain an adult's permission to participate in the trial.
  Parental Permission Required: Consent requirement where the participant is required to obtain their parent's permission to participate in the trial.
Period: Overall Study
Arm/Group | Adolescents: Consent Condition 1 | Adolescents: Consent Condition 2 | Adolescents: Consent Condition 3 | Parents: Consent Conditions 1-3
Started | 43 | 45 | 41 | 125
Completed | 43 | 45 | 41 | 125
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All parent participants are considered one study arm as they were not randomized to just one of the three consent conditions (as the adolescent participants were), but rather were presented with information on all 3 consent conditions and commented on the acceptability of each.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adolescents: Consent Condition 1 | Adolescents: Consent Condition 2 | Adolescents: Consent Condition 3 | Parents: Consent Conditions 1-3 | Total
Number analyzed (Participants) | 43 | 45 | 41 | 125 | 254
Age, Customized [Count of Participants; unit: Participants]
  14 years old | 1 | 1 | 0 | 0 | 2
  15 years old | 7 | 3 | 5 | 0 | 15
  16 years old | 11 | 8 | 15 | 0 | 34
  17 years old | 24 | 33 | 21 | 0 | 78
  >= 18 years old | 0 | 0 | 0 | 125 | 125
Sex: Female, Male [Count of Participants; unit: Participants] — sex assigned at birth
  Participants
    Female | 23 | 24 | 22 | 63 | 132
    Male | 20 | 21 | 19 | 62 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 8 | 18 | 48
  Not Hispanic or Latino | 30 | 33 | 32 | 103 | 198
  Unknown or Not Reported | 2 | 1 | 1 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 0 | 3 | 6
  Asian | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 0 | 2
  Black or African American | 19 | 27 | 21 | 73 | 140
  White | 9 | 7 | 14 | 31 | 61
  More than one race | 7 | 6 | 5 | 8 | 26
  Unknown or Not Reported | 5 | 3 | 0 | 10 | 18
Gender Identity [Count of Participants; unit: Participants] — Population: Gender identity data was not collected on Parent participants.
  Participants
    number analyzed (Participants) | 43 | 45 | 41 | 0 | 129
    Woman | 22 | 24 | 23 |  | 69
    Gender queer or gender non-conforming | 0 | 1 | 0 |  | 1
    Man | 15 | 18 | 14 |  | 47
    Trans woman | 3 | 1 | 4 |  | 8
    Trans man | 2 | 0 | 0 |  | 2
    Other | 1 | 1 | 0 |  | 2
Sexual orientation [Count of Participants; unit: Participants] — Population: sexual orientation data was not collected on parent participants
  Participants
    number analyzed (Participants) | 43 | 45 | 41 | 0 | 129
    Bisexual | 11 | 11 | 11 |  | 33
    Gay, queer, or same gender loving | 12 | 15 | 9 |  | 36
    Straight or heterosexual | 18 | 17 | 19 |  | 54
    Questioning | 0 | 1 | 0 |  | 1
    Other | 2 | 1 | 2 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Mean Adolescent WTP Scores
Description: Comparing mean adolescent Willingness to Participate (WTP) scores across the three consent conditions and two trial types.
  WTP scores are based on the response to the question: "If offered the chance, how likely would you be to participate in the study?" Responses are collected using a Likert scale (definitely not participate, probably not participate, might or might not participate, probably participate, definitely participate) and converted to a numeric score with values ranging from 1 (definitely not participate) to 5 (definitely participate) for analysis.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Adolescents: Consent Condition 1: Autonomous minor consent
  Autonomous consent: Consent requirement where the participant is not required to get anyone's permission to participate in the trial.
Arm/Group | Adolescents: Consent Condition 1 | Adolescents: Consent Condition 2 | Adolescents: Consent Condition 3
Number analyzed (Participants) | 43 | 45 | 41
score on a scale | 3.7 (0.8) | 3.7 (1.2) | 3.5 (0.8)
Statistical Analysis 1: Comparison: Adolescents: Consent Condition 1 vs Adolescents: Consent Condition 2 vs Adolescents: Consent Condition 3; Test type: Superiority; p = 0.5148, Regression, Linear; Cohen's f square = 0.011, 95% CI 2-sided [0.001 to 0.101], Standard Error of Mean 0.208

2. Primary Outcome: Mean Parent WTS Scores
Description: Comparing mean parent Willingness to Support (WTS) scores across the three consent conditions and two trial types.
  WTS scores are based on the response to the question: "This is an acceptable approach to consent for your teenager's participation in the study." Responses are collected using a Likert scale (strongly disagree, disagree, neither disagree nor agree, agree, strongly agree) and converted to a numeric score with values ranging from 1 (strongly disagree) to 5 (strongly agree) for analysis.
Time Frame: Day 1
Population: All parent participants commented on their Willingness to Support (WTS) each of the three consent conditions (autonomous minor consent, adult permission required, and parental permission required). For this reason, the Number Analyzed in each row of the table equals the total number of parent participants for the study (n=125)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents: Consent Conditions 1-3
Number analyzed (Participants) | 125
score on a scale
  Parent Consent Condition 1: Autonomous minor consent | 2.6 (1.5)
  Parent Consent Condition 2: Adult permission required | 3.1 (1.5)
  Parent Consent Condition 3: Parental permission required | 4.4 (1.0)
Statistical Analysis 1: Comparison: Parents: Consent Conditions 1-3; Test type: Superiority; p < .0001, Regression, Linear; Cohen's f square = 0.306, 95% CI 2-sided [0.169 to 0.389], Standard Error of Mean 0.149

3. Primary Outcome: Effects of the Study Agent (Stage of Development and Method of Delivery) on High-risk Minor Adolescents' WTP Scores
Description: This data reflects adolescent Willingness to Participate (WTP) scores by study agent/trial type. After review of hypothetical consent documents for 2 study agents in different stages of development and with different methods of delivery (based on real-world studies ATN 113 and HPTN 077), adolescents are asked "If offered the chance, how likely would you be to participate in the study?" Responses are collected using a Likert scale (definitely not participate, probably not participate, might or might not participate, probably participate, definitely participate) and converted to a numeric score with values ranging from 1 (definitely not participate) to 5 (definitely participate) for analysis.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adolescents: Consent Condition 1 | Adolescents: Consent Condition 2 | Adolescents: Consent Condition 3
Number analyzed (Participants) | 43 | 45 | 41
score on a scale
  Study agent 1 - ATN 113 | 3.6 (1.1) | 3.7 (1.3) | 3.6 (0.9)
  Study agent 2 - HPTN 077 | 3.8 (0.9) | 3.8 (1.2) | 3.4 (1.0)
Statistical Analysis 1: Comparison: Adolescents: Consent Condition 1 vs Adolescents: Consent Condition 2 vs Adolescents: Consent Condition 3; Test type: Superiority; p = 0.4324, GEE Linear model; Cohen's f square = 0.008, 95% CI 2-sided [0.001 to 0.073], Standard Error of Mean 0.213

4. Primary Outcome: Effects of the Study Agent (Stage of Development and Method of Delivery) on Parents' Acceptability Scores
Description: After review of hypothetical consent documents for 2 study agents in different stages of development and with different methods of delivery (based on real-world trials ATN 113 and HPTN 077), parents are presented with vignettes for the 3 different consent conditions (autonomous minor consent, adult permission required, parental permission required) and asked "How acceptable is this approach to research consent?". Responses are collected on a Likert scale (completely unacceptable, unacceptable, neither unacceptable not acceptable, acceptable, completely acceptable) and converted to a numeric score with values ranging from 1 (definitely not acceptable) to 5 (definitely acceptable) for analysis.
Time Frame: Day 1
Population: All parent participants commented on their Willingness to Support (WTS) each of the three consent conditions for each of the 2 trial types. For this reason, the Number Analyzed in each row of this data table equals the total number of parent participants for the study (n=125) as they all answered WTS for each.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parents: Consent Conditions 1-3
Number analyzed (Participants) | 125
score on a scale
  Autonomous minor consent study agent ATN 113 | 2.7 (1.6)
  Adult permission required study agent ATN 113 | 3.1 (1.6)
  Parental permission required study agent ATN 113 | 4.3 (1.2)
  Autonomous minor consent study agent HPTN 077 | 2.6 (1.5)
  Adult permission required study agent HPTN 077 | 3.1 (1.6)
  Parental permission required study agent HPTN 077 | 4.4 (1.1)
Statistical Analysis 1: Comparison: Parents: Consent Conditions 1-3; Test type: Superiority; p < .0001, GEE Linear model; Cohen's f square = 0.260, 95% CI 2-sided [0.175 to 0.374], Standard Error of Mean 0.149

ADVERSE EVENTS:
Time Frame: Adverse event data were collected on all participants during their one-time study visit
Description: All parent participants are considered one study 'arm' as they were not randomized to just one of the three consent conditions (as the adolescent participants were), but rather were presented with information on all 3 consent conditions and commented on the acceptability of each.
Arm/Group | Adolescents: Consent Condition 1 | Adolescents: Consent Condition 2 | Adolescents: Consent Condition 3 | Parents: Consent Conditions 1-3
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/45 | 0/41 | 0/125
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/45 | 0/41 | 0/125
Other Adverse Events (participants affected / at risk) | 0/43 | 0/45 | 0/41 | 0/125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/54/NCT03242954/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-10-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03242954/Prot_SAP_001.pdf